CLINICAL TRIAL: NCT06516224
Title: Evaluation of the Efficacy of the Anti-pigmenting Effect of a Routine of Facial Products in Subjects With Melasma
Brief Title: Anti-pigmenting Effect of a Routine of Facial Products in Subjects With Melasma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCY23-001
Record Dates: First submitted 2024-05-07; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Melasma
Keywords: melasma; hyperpigmentation
MeSH Terms: conditions — Melanosis; Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: single-center, randomised, 3 group study
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomized in three groups and will be treated differently taking into account only the original Melasma Area Severity Index (MASI) score at baseline:
  • An adaptive randomization scheme (minimization method) will be used to determine the treatment group (among the 3 available) to which eligible subjects will be enrolled in. This strategy will ensure a balance between treatment groups for one important prognostic factor, identified as 'baseline MASI'. When a new subject is eligible for randomization, the algorithm verifies the average MASI of the subjects in each group. The new subject will be allocated to a group in such a way that the imbalance is minimized among the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): dermocosmetic regimen consisting in Liftactiv(® B3 serum + Liftactiv® B3 retinol night cream (all Vichy Laboratoires, France) for 6 months + Mineral 89 cream + Sunscreen UVAage Inter SPF 50+
  Interventions: Other: Liftactiv® B3 Serum; Other: Liftactiv® B3 retinol night cream; Other: Sunscreen UVAage® Inter SPF 50+; Other: Mineral 89 cream
- Group 2 (Active Comparator): hydroquinone 4% (HQ4%, Hydroquinona 40 mg/g, Germed, Brazil) for 3 months followed by the dermocosmetic regimen (Liftactiv(® B3 serum + Liftactiv® B3 retinol night cream + Mineral 89 cream + Sunscreen UVAage Inter SPF 50+) for 3 months
  Interventions: Other: Liftactiv® B3 Serum; Other: Liftactiv® B3 retinol night cream; Other: Sunscreen UVAage® Inter SPF 50+; Other: Mineral 89 cream
- Group 3 (Active Comparator): Combination of hydroquinone, resorcinol corticosteroid (Kligman Trio, Vitacid Plus Cream, Claredor Brazil) for 3 months followed by the dermocosmetic regimen (Liftactiv(® B3 serum + Liftactiv® B3 retinol night cream + Mineral 89 cream + Sunscreen UVAage Inter SPF 50+) for 3 months
  Interventions: Other: Liftactiv® B3 Serum; Other: Liftactiv® B3 retinol night cream; Other: Sunscreen UVAage® Inter SPF 50+; Other: Mineral 89 cream

INTERVENTIONS:
Other: Liftactiv® B3 Serum — In Group 1: Application once daily for 6 months, 3-4 drops twice a day (morning before the sunscreen and evening) In Group 2 and Group 3: Application once daily, 3-4 drops twice a day (morning before the sunscreen and evening) for 3 months following HQ4% or Kligman Trio treatment.
Other: Liftactiv® B3 retinol night cream — In Group 1: Application once daily (morning) for 6 months In Group 2 and Group 3: During week 1, apply 2 evenings/week. During week 2, apply every other evening. During week 3, apply every evening. During nights when retinol night cream is not applied, replace with Mineral 89 cream for 3 months following HQ4% or Kligman Trio treatment.
Other: Sunscreen UVAage® Inter SPF 50+ — twice daily (morning and beginning of the afternoon)
Other: Mineral 89 cream — 2 drops in the morning before sunscreen application for 6 months

SUMMARY:
This 6 month, comparative study assesses the benefit of a dermocosmetic regimen (Serum B3 + B3 retinol night cream) for 6 months compared to hydroquinone 4% (the gold standard in hyperpigmentation) followed by the dermocosmetic regimen for 3 months or the Kligman Trio for 3 months followed by the dermocosmetic regimen for 3 months in adult women with melasma on the face.

DETAILED DESCRIPTION:
Study objective

1. Assessing the antipigmenting efficacy of the routine (serum B3 + B3 retinol night cream) in women with melasma.
2. Evaluation of Kligman Trio (KT) (Vitacid Plus) compared to the routine (serum B3 + B3 retinol night cream)
3. Evaluation of Hydroquinone 4% (HQ 4%) compared to the routine (serum B3 + B3 retinol night cream).
4. Assessment of the routine maintenance with SERUM B3 + retinol B3 night cream after 3 months of use of Klingman Trio (KT)(Vitacid plus) and HQ4%

Primary endpoint:

o Improvement of mMASI and MASI

Secondary endpoints:

* Improvement of Physician Global Assessment IGA for melasma
* Improvements on clinical parameters such as fine lines, skin tone, radiance, skin texture and skin elasticity evaluated by the investigator.
* Global efficacy by the subject and by the investigator (Physician's Global assessment)
* Global tolerance
* Safety
* Cosmetic acceptability
* Improvement of Quality of life (MelasQOL)
* Exposome questionnaire
* Questionnaire on hormonal status
* Improvement of the morphological and structural characteristics of ageing skin - By confocal microscopy (15 subjects per subgroup)
* Clinical scoring: hyperpigmentation scale
* Standard facial pictures with Colorface®
* Chromameter® measurements (target lesion assessment compared to non lesional surrounding skin)
* Tewameter® measurements
* Corneometer® measurements

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Phototype II-V
* 50% with sensitive skin (declarative);
* Subjects should be affected by well defined symmetrical (on both sides of the face) epidermal melasma (clinically diagnosed under Wood's light examination) lasting since more than a year

Exclusion Criteria:

* Subjects under topical or systemic retinoids;
* Subjects having used topical tretinoin within 3 months or topical hydroquinone within 6 months prior to inclusion;
* Subjects under systemic immunosuppressants and considered immune compromised
* Subjects under active treatment of melasma (including topicals or procedures) within the last 3 months
* Pregnant women and/or breastfeeding women
* Subjects with a recent change in contraception (since less than 6 months);
* Subjects known allergy to any component of tested product;
* Subjects not presenting with the conditions needed to comply with the protocol;
* Subjects without any other dermatological conditions on the face
* Subject under menopause phase with hormonal replace therapy
* Subjects in the initial phase, change or discontinuation of hormonal treatment (estroprogesterone, cyproteron acetate, androgenic...) in the last 3 months;
* Subjects currently using any medication, which in the opinion of the investigator, may affect the evaluation of the study product, or place the subject at undue risk.
* Subjects unable to give their informed consent.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
antipigmenting assessment | Day 84
  Melasma Area Severity Index (MASI)
antipigmenting assessment | Day 84
  modified Melasma Area Severity Index (mMASI)
antipigmenting assessment | Day 168
  Melasma Area Severity Index(MASI)
antipigmenting assessment | Day 168
  modified Melasma Area Severity Index (mMASI)

SECONDARY OUTCOMES:
antipigmenting assessment | Day-28
  Melasma Area Severity Index(MASI)
antipigmenting assessment | Day-28
  modified Melasma Area Severity Index (mMASI)
antipigmenting assessment | baseline
  Melasma Area Severity Index(MASI)
antipigmenting assessment | baseline
  modified Melasma Area Severity Index (mMASI)
antipigmenting assessment | Day 28
  Melasma Area Severity Index(MASI)
antipigmenting assessment | Day 28
  modified Melasma Area Severity Index (mMASI)
antipigmenting assessment | Day 56
  Melasma Area Severity Index(MASI)
antipigmenting assessment | Day 56
  modified Melasma Area Severity Index (mMASI)
antipigmenting assessment | Day 112
  Melasma Area Severity Index(MASI)
antipigmenting assessment | Day 112
  modified Melasma Area Severity Index (mMASI)
antipigmenting assessment | Day 140
  Melasma Area Severity Index(MASI)
antipigmenting assessment | Day 140
  modified Melasma Area Severity Index (mMASI)
Investigator Global Assessment (IGA) assessment | Day -28
  IGA score
Investigator Global Assessment (IGA) assessment | baseline
  IGA score
Investigator Global Assessment (IGA) assessment | Day 28
  IGA score
Investigator Global Assessment (IGA) assessment | Day 56
  IGA score
Investigator Global Assessment (IGA) assessment | Day 84
  IGA score
Investigator Global Assessment (IGA) assessment | Day 112
  IGA score
Investigator Global Assessment (IGA) assessment | Day 140
  IGA score
Investigator Global Assessment (IGA) assessment | Day 168
  IGA score
Clinical assessment (fine lines, skin tone, radiance, texture and elasticity) | Day -28
  scores 0 to 5
Clinical assessment (fine lines, skin tone, radiance, texture and elasticity) | baseline
  scores 0 to 5
Clinical assessment (fine lines, skin tone, radiance, texture and elasticity) | Day 28
  scores 0 to 5
Clinical assessment (fine lines, skin tone, radiance, texture and elasticity) | Day 84
  scores 0 to 5
Clinical assessment (fine lines, skin tone, radiance, texture and elasticity) | Day 168
  scores 0 to 5
Clinical scoring hyperpigmentation | baseline
  scale 0 to 10
Clinical scoring hyperpigmentation | Day 28
  scale 0 to 10
Clinical scoring hyperpigmentation | Day 56
  scale 0 to 10
Clinical scoring hyperpigmentation | Day 84
  scale 0 to 10
Clinical scoring hyperpigmentation | Day 112
  scale 0 to 10
Clinical scoring hyperpigmentation | Day 140
  scale 0 to 10
Clinical scoring hyperpigmentation | Day 168
  scale 0 to 10
Clinical scoring target lesion comparing to surrounding skin | baseline
  scale 0 to 10
Clinical scoring target lesion comparing to surrounding skin | Day 28
  scale 0 to 10
Clinical scoring target lesion comparing to surrounding skin | Day 56
  scale 0 to 10
Clinical scoring target lesion comparing to surrounding skin | Day 84
  scale 0 to 10
Clinical scoring target lesion comparing to surrounding skin | Day 112
  scale 0 to 10
Clinical scoring target lesion comparing to surrounding skin | Day 140
  scale 0 to 10
Clinical scoring target lesion comparing to surrounding skin | Day 168
  scale 0 to 10
Subject global efficay rating | Day 28
  rating
Subject global efficay rating | Day 56
  rating
Subject global efficay rating | Day 84
  rating
Subject global efficay rating | Day 112
  rating
Subject global efficay rating | Day 140
  rating
Subject global efficay rating | Day 168
  rating
Investigator global efficay rating | Day 28
  rating
Investigator global efficay rating | Day 56
  rating
Investigator global efficay rating | Day 84
  rating
Investigator global efficay rating | Day 112
  rating
Investigator global efficay rating | Day 140
  rating
Investigator global efficay rating | Day 168
  rating
Cosmetic acceptability | Day 28
  questionnaire
Cosmetic acceptability | Day 56
  questionnaire
Cosmetic acceptability | Day 84
  questionnaire
Cosmetic acceptability | Day 112
  questionnaire
Cosmetic acceptability | Day 140
  questionnaire
Cosmetic acceptability | Day 168
  questionnaire
Evolution of quality of life | Day -28
  MelasQoL
Evolution of quality of life | baseline
  MelasQoL
Evolution of quality of life | Day 28
  MelasQoL
Evolution of quality of life | Day 56
  MelasQoL
Evolution of quality of life | Day 84
  MelasQoL
Evolution of quality of life | Day 112
  MelasQoL
Evolution of quality of life | Day 140
  MelasQoL
Evolution of quality of life | Day 156
  MelasQoL
images | baseline
  Standard facial pictures with Colorface® using standard 60, cross polarized, UV and no filters lights.
images | Day 28
  Standard facial pictures with Colorface® using standard 60, cross polarized, UV and no filters lights.
images | Day 56
  Standard facial pictures with Colorface® using standard 60, cross polarized, UV and no filters lights.
images | Day 84
  Standard facial pictures with Colorface® using standard 60, cross polarized, UV and no filters lights.
images | Day 112
  Standard facial pictures with Colorface® using standard 60, cross polarized, UV and no filters lights.
images | Day 140
  Standard facial pictures with Colorface® using standard 60, cross polarized, UV and no filters lights.
images | Day 168
  Standard facial pictures with Colorface® using standard 60, cross polarized, UV and no filters lights.
Skin quality | baseline
  Chromameter, Individual Typology Angle (ITA)
Skin quality | Day 28
  Chromameter, Individual Typology Angle (ITA)
Skin quality | Day 56
  Chromameter, Individual Typology Angle (ITA)
Skin quality | Day 84
  Chromameter, Individual Typology Angle (ITA)
Skin quality | Day 112
  Chromameter, Individual Typology Angle (ITA)
Skin quality | Day 140
  Chromameter, Individual Typology Angle (ITA)
Skin quality | Day 168
  Chromameter, Individual Typology Angle (ITA)
transepidermal water loss | baseline
  Tewameter
transepidermal water loss | Day 28
  Tewameter
transepidermal water loss | Day 56
  Tewameter
transepidermal water loss | Day 84
  Tewameter
transepidermal water loss | Day 112
  Tewameter
transepidermal water loss | Day 140
  Tewameter
transepidermal water loss | Day 168
  Tewameter
skin hydration | baseline
  Corneometer
skin hydration | Day 28
  Corneometer
skin hydration | Day 56
  Corneometer
skin hydration | Day 84
  Corneometer
skin hydration | Day 112
  Corneometer
skin hydration | Day 140
  Corneometer
skin hydration | Day 168
  Corneometer
confocal | baseline
  confocal measurements (15 subjects)
confocal | Day 84
  confocal measurements (15 subjects)
confocal | Day 168
  confocal measurements (15 subjects)
exposome questionnaire | baseline
  questionnaire
Melasma status | baseline
  questionnaire
adverse events | baseline
  reporting
adverse events | Day 28
  reporting
adverse events | Day 56
  reporting
adverse events | Day 84
  reporting
adverse events | Day 112
  reporting
adverse events | Day 140
  reporting
adverse events | Day 168
  reporting

CONTACTS AND LOCATIONS:
Overall Officials: Claire Deloche-Bensmain, PhD, Study Director — La Roche Posayl Laboratoires Dermatologiques
Locations (1):
- CIDP, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
the protocol will be shared by the sponsor upon reasonable request for one year after the end of the study
Supporting Information: Study Protocol
Time Frame: one after finishing study
Access Criteria: upon request to the sponsor